CLINICAL TRIAL: NCT01882335
Title: Saving Brains In Uganda And Burkina Faso (PROMISE Saving Brains)
Brief Title: Saving Brain in Uganda and Burkina Faso
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Makerere University (Other)
Collaborators: Centre Muraz (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Grant # 0064-03; Grant # 0064-03 (Other: GRAND CHALLENGES CANADA)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-04

CONDITIONS: Poor Performance Status; Neurologic Deficits; Mixed Behavior and Emotional Disorder; Malnutrition; Infections, Hospital
Keywords: Human capital formation
MeSH Terms: conditions — Neurologic Manifestations; Malnutrition; Cross Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral (Experimental): Peer support for mothers to encourage them to exclusively breastfeed their babies for 6 months
  Interventions: Behavioral: Peer support for exclusive breastfeeding
- Control (No Intervention): No peer support for exclusive breastfeeding

INTERVENTIONS:
Behavioral: Peer support for exclusive breastfeeding — Pregnant women were identified and randomized to peer support for exclusive breastfeeding in clusters. They were followed up for 6 months post delivery.
  Other Names: Peer support
  Arms: Behavioral

SUMMARY:
The study will estimate the effect of peer-counseling for exclusive breast feeding (EBF) in the first 6 months of life on cognition and other determinants of human capital formation including behavioral and emotional status; school readiness and attainment; health status; fine and gross motor skills; physical growth; and household economic status.

DETAILED DESCRIPTION:
Between 2006 and 2008 we carried out a cluster randomized study (PROMISE-EBF) to establish the effect of individual home based peer counselling on exclusive breast feeding (EBF). The results, published in the Lancet in 2011 were remarkable(Tylleskar T, et al). The PROMISE-EBF trial which compared mothers in the intervention arm that were offered at least 5 peer-visits promoting EBF to mothers in the control arm, that received the standard of care showed a doubling in the prevalence of EBF in the intervention arm. Community-based peer counsellors increased the EBF rate in Uganda and Burkina Faso from about 40% to 80%.

The current study will trace and re-enrol at least 70% of the children involved in the PROMISE-EBF study. These children are now aged between 5 and 7 years.

The primary objective of the current study is to evaluate the effect of peer-counselling for EBF in the first six months of life on human capital formation among children in Uganda and Burkina Faso.

This study will contribute to a crucial wider discussion on external validity regarding the relationship between EBF and intellectual performance and mental health. In the social area, this study will identify solutions to potential barriers that limit scale up for peer-counselling for EBF. From the business perspective, the study will identify the best business model for affordable, acceptable and cost effective ways of delivering peer counselling for EBF in Burkina Faso and Uganda. If this intervention is found effective, and is adopted, it could improve productivity in adulthood and work towards breaking the cycle of poverty.

ELIGIBILITY:
Inclusion Criteria:

* Children whose mothers participated in the original intervention of peer support for exclusive breastfeeding (EBF).
* Informed caregiver consent

Exclusion Criteria:

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | one year
  Proportion of children with impaired cognitive function in intervention compared to the control group

SECONDARY OUTCOMES:
Cost-effectiveness of promoting peer-counselling for exclusive breastfeeding in the first six months of life to support human capital formation | 3 months
  Determine the cost of promoting peer counselling for exclusive breastfeeding in relation to the cost of attending to children with poor outcomes

OTHER OUTCOMES:
School attainment | One year
  School attainment in the intervention compared to school attainment in the control group
School readiness | One year
  The age at which children are ready to start school in the intervention compared to the control group.
Physical growth | One year
  Compare the proportion of children with poor nutritional status in the intervention and control group.
Behavioural and emotional status | One year
  Behavioral and emotional status of children in the intervention compared to those in the control group
Household economic status | One year
  Assess the social economic status in the intervention compared to the social economic status in the control group.
Motor skills | One year
  Compare motor skills of children in the intervention compared to the control group using MABC

CONTACTS AND LOCATIONS:
Overall Officials: James K Tumwine, PhD, Principal Investigator — Makerere University
Locations (1):
- Makerere University, Kampala, Uganda

REFERENCES:
- [Derived] Engebretsen IMS, Nalugya JS, Skylstad V, Ndeezi G, Akol A, Babirye JN, Nankabirwa V, Tumwine JK. "I feel good when I drink"-detecting childhood-onset alcohol abuse and dependence in a Ugandan community trial cohort. Child Adolesc Psychiatry Ment Health. 2020 Oct 24;14:42. doi: 10.1186/s13034-020-00349-z. eCollection 2020. PMID 33110445
- [Derived] Tumwine JK, Nankabirwa V, Diallo HA, Engebretsen IMS, Ndeezi G, Bangirana P, Sanou AS, Kashala-Abotnes E, Boivin M, Giordani B, Elgen IB, Holding P, Kakooza-Mwesige A, Skylstad V, Nalugya J, Tylleskar T, Meda N. Exclusive breastfeeding promotion and neuropsychological outcomes in 5-8 year old children from Uganda and Burkina Faso: Results from the PROMISE EBF cluster randomized trial. PLoS One. 2018 Feb 23;13(2):e0191001. doi: 10.1371/journal.pone.0191001. eCollection 2018. PMID 29474479